CLINICAL TRIAL: NCT02727699
Title: XanADu: A Phase II, Double-Blind, 12-Week, Randomised, Placebo-Controlled Study to Assess the Safety, Tolerability and Efficacy of Xanamem™ in Subjects With Mild Dementia Due to Alzheimer's Disease (AD)
Brief Title: A Phase II Study to Assess the Safety, Tolerability and Efficacy of Xanamem™ in Subjects With Mild Dementia Due to AD (XanADu)
Acronym: XanADu
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actinogen Medical (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACW0002
Record Dates: First submitted 2016-03-21; First posted 2016-04-05 (Estimated); Results first posted 2021-05-06 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2022-04

CONDITIONS: Dementia, Alzheimer Type
Keywords: Dementia; Alzheimer's Disease; Xanamem; UE2343 (Laboratory Code for Xanamem); Cortisol; XanADu; Actinogen; 11β-HSD1; 11-beta-Hydroxysteroid Dehydrogenase Type 1; Mild Alzheimer's Disease; Cognitive Impairments; emestedastat
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction | interventions — UE2343

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Xanamem™ (Experimental): Oral Xanamem™ capsules 10mg, to be administered once daily
  Interventions: Drug: Xanamem™
- Placebo (Placebo Comparator): Matching placebo which is identical in appearance to the test product except that it contains no active ingredient, to be administered once daily
  Interventions: Drug: Placebo (for Xanamem™)

INTERVENTIONS:
Drug: Xanamem™ — Xanamem™ is formulated in green and cream coloured size 3, Coni-Snap shaped gelatin capsules as an excipient blend at a dose of 10mg. It contains active pharmaceutical ingredient of UE2343
  Other Names: UE2343
  Arms: Xanamem™
Drug: Placebo (for Xanamem™) — Excipient blend capsules manufactured to mimic Xanamem™ capsules
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This XanADu Phase II study in mild Alzheimer's Disease (AD) is to assess the safety, tolerability and efficacy of Xanamem in subjects with mild dementia due to Alzheimer's Disease. Subjects will be randomized to receive either 10mg once daily Xanamem or Placebo at a 1:1 ratio in a double-blinded fashion.

DETAILED DESCRIPTION:
This is a Phase II, randomised, multi-centre, double-blind, placebo-controlled proof-of-concept study to assess the safety, tolerability and efficacy of oral Xanamem once daily in adult subjects with mild dementia due to AD.

Based on Xanamem's mode of action on hippocampal function, amnestic symptoms may respond best, thus favouring the inclusion of mild dementia due to AD, with given evidence of disease progression. Subjects will be treated in a double-blind fashion, where both the investigators and subjects will be unaware of the treatment assignments, to minimise any subjective or unrecognised bias carried by the investigators and subjects. Placebo will be used as the comparator in this study.

It is planned to randomise approximately 174 subjects at approximately 25 study sites in three countries (Australia, United Kingdom, and United States), with the aim to enrol 7 to 10 subjects at each study site. Subject enrolment will be competitive but a cap of 20 subjects per study site is to be established to avoid any side effects. In case the sample composition at one study site is creating concerns, an enrolment stop can also occur at fewer than 20 subjects.

At study end, a total of 185 subjects were randomised into this study and received active treatment.

The data safety monitoring board (DSMB) will periodically meet for the review of accumulating safety study data and will also be involved in the interim analysis.

At the Baseline visit (Week 0), eligible subjects will be randomised on a 1:1 ratio to receive either Xanamem administered orally once daily (QD) for the treatment group or matching placebo for the placebo group. Subjects will return to the study site for visits at Week 4 and Week 8, End of Treatment (Week 12) and Follow-up (4 weeks post last dose of study drug) visits, at which study assessments will be performed.

Ad hoc telephone contact may also occur at any other time-point throughout the study, if deemed necessary by the investigator/study nurse, or if the subject wishes to report an Adverse Event (AE)

Subjects will be interviewed and examined at the study site at each visit and will complete a variety of questionnaires and routine safety evaluations.

Optional Pharmacodynamic (PD) sampling will be performed at specific visits. Subjects who do not provide consent for this optional sub-study will still be eligible for the main study.

The overall study duration for an individual subject will be 17 to 20 weeks, including a screening period of one to 4 weeks, a double-blind treatment period of 12 weeks, and a follow-up period of 4 weeks. The total duration of the study is expected to be 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 50 years or older at the time of informed consent.
2. Female Subjects:

   1. Post menopausal women, defined as no menses for 12 months without an alternative medical cause. If there is any concern about the menopausal status of a prospective female subject, a follicle stimulating hormone test (FSH) should be requested to confirm post-menopausal status. Post menopausal women confirmed by FSH level > 40 mIU (milli-international units per milliliter) /mL, will be confirmed by central laboratory.
   2. Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and Baseline, and be willing to use highly effective methods of contraception from the Screening visit until 3 months after last dose of study drug. If re-test is required, a local urine pregnancy test will be performed at Baseline to determine if the subject can continue to randomisation.
   3. Are permanently sterile or have had a hysterectomy, bilateral salpingectomy or bilateral oophorectomy.
   4. Women must not be breastfeeding.
3. Male Subjects:

   1. Who are sexually active, fertile men must use highly effective methods of contraception from Day 1 until 3 months after last dose of study drug if their partners are WOCBP.
   2. Who are permanently sterile or have had bilateral orchiectomy.
4. Diagnosis of mild dementia due to Alzheimer's disease (AD) with increased level of certainty (provided by evidence of clinical deterioration within the 6 months preceding Screening, as assessed by the investigator) as determined by the National Institute of Ageing (NIA) and the Alzheimer's Association (AA) workgroup.
5. Mild dementia due to probable AD with Mini-Mental Status Examination (MMSE) 20 to 26 (inclusive).
6. Clinical Dementia Rating Scale (CDR) Global Score of 0.5 to 1.0.
7. A brain magnetic resonance imaging (MRI) or computed tomography (CT) scan in the 12 months preceding Screening that in the investigator's opinion is consistent with AD as the principle aetiology of the dementia with no other clinically significant abnormality, e.g. another principle underlying aetiology of the subject's dementia, or a lesion which could affect cognition e.g. a brain tumour or large stroke.
8. On stable dose of acetylcholinesterase (AChEI) and/or memantine (at least 3 months prior to Screening) OR treatment-naïve. Initiating AChEIs or memantine during the study will not be permitted.
9. Apart from a clinical diagnosis of mild dementia due to AD, the subject must be in good health as determined by the investigator, based on medical history and screening assessments.
10. Has a consenting study partner who, in the investigator's judgement, has frequent and sufficient contact with the subject to be able to provide accurate information as to the subject's cognitive and functional abilities. The study partner must be available to provide information to the investigator and study site staff about the subject and agrees to attend all study site visits in person for scale completion. A study partner should be available for the duration of the study. The measure of adequate availability will be at the investigator's discretion.
11. Must be willing and able to comply with the requirements of the protocol and must be available to complete the study.
12. Must satisfy a medical examiner about their fitness to participate in the study.
13. Must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Clinically significant abnormalities in vital signs (blood pressure, heart rate, respiration rate and oral temperature), as determined by the investigator.
2. Clinically significant abnormal haematology, biochemistry and urine examination values, specifically abnormal liver and renal function and Vitamin B12 levels below lower threshold since these parameters may impact cognitive function, as determined by the investigator.
3. Has had a significant systematic illness or infection within the past 4 weeks prior to randomisation, as determined by the investigator.
4. Clinically significant neurological disease other than AD, such as (but not limited to) Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumour, progressive supranuclear palsy, seizure disorder, subdural haematoma, multiple sclerosis or a history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.
5. Subjects with clinical evidence of peripheral neuropathy or historical evidence of clinically significant nerve conduction abnormalities.
6. Has had a stroke within the year prior to randomisation, as determined by the investigator.
7. Has a lifetime diagnosis of a major psychiatric disorder (other than dementia), based on the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition criteria. This includes but is not limited to schizophrenia, schizoaffective disorder, bipolar affective disorder, alcohol dependence syndrome or major depressive disorder.
8. Has a history of disease directly related to the hypothalamus, the pituitary and/or the adrenal glands which affect the hypothalamic-pituitary-adrenal axis function.
9. Has uncontrolled clinical conditions relating to glucose and lipid metabolism.
10. Clinically significant electrocardiogram (ECG) abnormalities, including Corrected QT interval (QTc) > 450 ms, following ECG tracings at Screening.
11. Use of any prohibited medication as detailed in the study protocol.
12. Participation in another clinical study of an investigational drug or device whereby the last investigational drug/device administration is within 60 days of Screening.
13. Inability to communicate well with the investigator (i.e. language problem, non-fluent English [as scales will be provided in English only], poor mental development or impaired cerebral function).
14. Subject will undergo the tests, Alzheimer's Disease Assessment Scales (ADAS)-Cog v14, CDR-Sum of Boxes (SOB), MMSE, Neuropsychological Test Battery (NTB; executive domain) and RAVLT at the indicated time-points to avoid uncontrolled learning effects. Subjects who need to perform these tests externally to and in parallel with this study will be excluded.
15. Subject has ingested any food or drink containing grapefruit, Seville oranges, star fruit or derived products (e.g. fruit juice), for at least 3 days prior to the first administration of study drug.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bill Ketelbey, MD, Study Chair — Actinogen Medical; Alan Boyd, MD, FFPM, Study Director — Actinogen Medical
Locations (25):
- United States (14):
  - Tucson Neuroscience Research, LLC, Tucson, Arizona
  - National Research Institute, Los Angeles, California
  - PCND Neuroscience Research Institute, Poway, California
  - Pacific Research Network, Inc., San Diego, California
  - Research Alliance Inc., Clearwater, Florida
  - The Neurology Research Group, LLC, Miami, Florida
  - Compass Research LLC, Orlando, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - NeuroStudies.Net, LLC, Decatur, Georgia
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - Richmond Behavioral Associates, Staten Island, New York
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - The Clinical Trial Center, Jenkintown, Pennsylvania
- Australia (5):
  - Central Coast Neurosciences Research, Central Coast, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - KaRa Institute of Neurological Diseases, Macquarie Park, New South Wales
  - Medical & Cognitive Research Unit, Heidelberg Repatriation Hospital - Austin Health, Heidelberg West, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
- United Kingdom (6):
  - The Research Institute for the Care of Older People, Bath, Combe Park
  - Manchester Mental Health & Social Care Trust - Dementia Research Office - Park House North Manchester General Hospital, Manchester, Lancashire
  - West London Mental Health Trust, Isleworth, London
  - St Pancras Clinical Research, Kings Cross, London
  - Institute of Clinical Sciences, Queen's University Belfast, Belfast, Northern Ireland
  - Centre for Clinical Brain Sciences, Centre for Dementia Prevention, The University of Edinburgh, Edinburgh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Webster SP, McBride A, Binnie M, Sooy K, Seckl JR, Andrew R, Pallin TD, Hunt HJ, Perrior TR, Ruffles VS, Ketelbey JW, Boyd A, Walker BR. Selection and early clinical evaluation of the brain-penetrant 11beta-hydroxysteroid dehydrogenase type 1 (11beta-HSD1) inhibitor UE2343 (Xanamem). Br J Pharmacol. 2017 Mar;174(5):396-408. doi: 10.1111/bph.13699. Epub 2017 Jan 25. PMID 28012176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited based on physician referral between March 2017 to November 2018 when enrolment completed. This was a global, multi-center study involving 27 study sites, of which, 24 sites had randomised subjects to the study.The study planned to enrol 7 to 10 subjects at each study site.
Pre-assignment Details: It was planned that approximately 174 subjects would be enrolled to ensure 156 subjects would complete the 12 week double-blind study period (78 subjects in each treatment group). At study-end, in total, 457 subjects were screened, of whom 185 subjects were randomised (91:94 Xanamem to placebo) to the study with 171 subjects completed.
Groups:
- Xanamem™: Oral Xanamem™ capsules 10mg, to be administered once daily
  Xanamem™: Xanamem™ is formulated in green and cream coloured size 3, Coni-Snap shaped gelatin capsules as an excipient blend at a dose of 10mg. It contains active pharmaceutical ingredient of UE2343 (Laboratory code for Xanamem)
Period: Overall Study
Arm/Group | Xanamem™ | Placebo
Started | 91 | 94
Completed | 82 | 89
Not Completed | 9 | 5
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: The FAS comprised all subjects randomised who received at least one dose of study drug and had at least one valid post-baseline measurement where changes from Baseline were analysed.
  Demographic data and subject characteristics at Baseline were summarised overall and by treatment, group using descriptive summary statistics for the Full Analysis Set (FAS) to include: age, gender and race. Baseline characteristic results of height, weight, BMI were also summarised overall and by treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Xanamem™ | Placebo | Total
Number analyzed (Participants) | 91 | 94 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 24 | 43
  >=65 years | 72 | 70 | 142
Age, Continuous [Median (Standard Deviation); unit: years] — Age was calculated as (informed consent year-birth year).
  years | 71.3 (8.71) | 70.8 (8.20) | 71.0 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 54 | 106
  Male | 39 | 40 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 13 | 30
  White | 65 | 74 | 139
  More than one race | NA — Data not available (NA) | NA — Data not available (NA) | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants] — Subject Allocation By Study Sites by Country Region
  participants
    United States | 53 | 55 | 108
    United Kingdom | 14 | 15 | 29
    Australia | 24 | 24 | 48
Height [Mean (Standard Deviation); unit: centimetres (cm)] — Population: Number of subjects in the specified category with non-missing values in the Full Analysis Set (FAS).
  centimetres (cm) | 165.49 (9.665) | 166.36 (8.964) | 165.94 (9.295)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram / square meter (kg/m^2)] — The overall mean (SD) Body Mass Index (BMI) of subjects was 27.19 (5.855) kg/m^2 and ranged from 17.9 kg/m^2 to 52.5 kg/m^2. Population: Baseline value is defined as the latest observation prior to or on the date of the first dose of study drug.
  kilogram / square meter (kg/m^2) | 27.31 (5.024) | 27.08 (6.570) | 27.19 (5.855)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 74.90 (15.964) | 74.88 (18.774) | 74.89 (17.424)

OUTCOME MEASURES:

1. Primary Outcome: ADAS-Cog v14
Description: Change in Alzheimer's Disease Assessment Scales - Cognitive Subscale Score, version 14 (ADAS-Cog v14) Total scores of ADAS Cog 14 range from 0 to 90, with higher scores indicating greater disease severity.
Time Frame: Baseline, Week 12
Population: The ADAS-cog v14 includes the following 14 items, with a Total scoring range of 0 - 90. Higher scores indicate greater disease severity
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Xanamem™ | Placebo
Number analyzed (Participants) | 86 | 92
units on a scale | -1.5 (6.47) | -0.7 (6.65)

2. Primary Outcome: AD COMposite Scores
Description: Change in AD COMposite Scores (ADCOMs- ADCOMs, composite score is derived from a weighted linear combination of items from commonly used outcome scales Cognitive Subscale Version 14 [ADAS-Cog v14], Clinical Dementia Rating Scale - Sum of Boxes [CDR-SOB], and Mini-Mental Status Examination [MMSE]. Th ADCOMs range: 0 - 1.97, whereas a lover score is interpreted as a better result.
  Included scales:
  ADAS-Cog v14 (range: 0-90): A lower score is indicative of better cognition, a higher score indicates higher cognitive impairment.
  CDR-SOB (range: 0-18): A lower score is indicative of better cognition, a higher score indicates higher cognitive impairment.
  MMSE (range: 0-30): A higher score is indicative of better cognition, a lower score indicates higher cognitive impairment.
Time Frame: Baseline, Week 12
Population: ADCOMs, composite score (0 - 1.97) is derived from ADAS-Cog v14, CDR-SOB, and MMSE. Analysis of Change from Baseline to Week 12/end of treatment (EOT) in ADCOMs from the Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xanamem™ | Placebo
Number analyzed (Participants) | 86 | 92
score on a scale | 0.02472 (0.144135) | 0.01908 (0.151502)

3. Secondary Outcome: RAVLT
Description: Change in Rey Auditory Verbal Learning Test (RAVLT) RAVLT will be administered using five trials, with individual scores from 0-15. The total score is the combined score of all five trials, ranging from 0 to 75, whereas a lower score is considered a worse outcome and a higher score a better outcome.
Time Frame: Baseline, Week 12
Population: Analysis of Change from Baseline to Week 12/EOT in RAVLT from the Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xanamem™ | Placebo
Number analyzed (Participants) | 86 | 92
score on a scale
  Recall List A - Total number of correct words: number analyzed (Participants) | 86 | 90
  Recall List A - Total number of correct words | 0.3 (6.54) | 0.4 (6.31)
  Recall List B - Number of correct words: number analyzed (Participants) | 86 | 90
  Recall List B - Number of correct words | 0.3 (1.63) | 0.1 (1.30)
  Final recall of List A - Number of correct words: number analyzed (Participants) | 85 | 90
  Final recall of List A - Number of correct words | 0.2 (3.14) | 0.4 (2.40)

4. Secondary Outcome: CDR-SOB
Description: Change in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SOB) The CDR is obtained through semi-structured interviews of patients and informants, and cognitive functioning is rated in six domains of functioning: memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care.
  Each domain is rated on a five-point scale of functioning as follows: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment.
  The CDR-SOB is based on summing each of the domain box scores, with scores ranging from 0-18, whereas lower scores represent better outcomes and higher scores worse outcomes.
Time Frame: Baseline, Week 12
Population: CDR-SOB score (0 - 18) is a sum of all six items of CDR-SOB. CDR-SOB score will be analysed for each visit as actual values and change from Baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xanamem™ | Placebo
Number analyzed (Participants) | 85 | 91
score on a scale | 0.25 (1.276) | 0.16 (1.325)

5. Secondary Outcome: MMSE
Description: Change in Mini-Mental Status Examination (MMSE) MMSE total score (0 - 30) is a sum of all 30 point questionnaire of MMSE. A score of 20 to 24 suggests mild dementia, 13 to 20 suggests moderate dementia, and less than 12 indicates severe dementia.
Time Frame: Baseline, Week 12
Population: MMSE is a 30 point questionnaire used to screen for dementia and to estimate the severity and progression of cognitive impairment. MMSE will be analysed for each visit as actual values and change from Baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xanamem™ | Placebo
Number analyzed (Participants) | 86 | 91
score on a scale | 0.2 (3.09) | -0.2 (2.85)

6. Secondary Outcome: NPI (Neuropsychiatric Inventory)
Description: Change in Neuropsychiatric Inventory (NPI) The NPI includes questions to ten behavioural and two neurodegenerative domains.
  Raters recorded neuropsychiatric symptoms using a 1-4 scale for frequency and a 1-3 scale for severity for each item in the instrument, with the score for each domain being: domain score = frequency x severity.
  The total score is calculated by adding the scores of the first 10 domain scores.
  The two neurodegenerative items are not included in the NPI total score as they form part of the depression syndrome in some patients and were specifically excluded from the dysphoria subscale of the NPI in order to allow that subscale to focus on mood symptoms.
  The total NPI-score minimum is 0 and the maximum 144. A lower score is considered a better outcome, a higher score a worse outcome.
Time Frame: Baseline, Week 12
Population: The NPI total score is calculated by multiplying the frequency and severity rates per domain (maximum score per domain is 12) and then calculating the total of all domains (total NPI-score minimum is 0 and maximum 144). Total distress score (0 - 60) will summarised descriptively. NPI total score will not be calculated if any sub item is missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Xanamem™ | Placebo
Number analyzed (Participants) | 85 | 92
units on a scale
  NPI Total Score | 0.9 (8.67) | 0.8 (9.09)
  Delusions | 0.0 (0.38) | 0.1 (0.87)
  Hallucinations | 0.1 (0.60) | 0.0 (0.36)
  Agitation/Aggression | 0.2 (2.02) | 0.2 (1.91)
  Depression/Dysphoria | 0.0 (1.34) | 0.0 (1.91)
  Anxiety | 0.1 (1.70) | -0.4 (2.08)
  Elation/Euphoria | 0.1 (0.92) | 0.0 (0.67)
  Apathy/Indifference | 0.0 (2.18) | 0.3 (2.11)
  Disinhibition | 0.1 (1.15) | 0.1 (1.03)
  Irritability/Lability | 0.1 (1.94) | 0.5 (2.17)
  Aberrant Motor Behavior | -0.1 (2.98) | 0.2 (2.37)
  Sleep | 0.2 (2.47) | 0.0 (1.83)
  Appetite and Eating Disorders | 0.1 (3.18) | -0.1 (2.02)

7. Secondary Outcome: NTB - Executive Domain
Description: Change in Neuropsychological Test Batteries (NTB) - Executive Domains: Controlled Oral Word Association - Test (COWAT) and Total Correct Response (CFT) Total NTB score is the sum of COWAT and CFT. During the COWAT test, the subject is asked to mention as many words as possible beginning with different letters (F, A, S) within 1 minute each. The number of words for each letter is recorded, the score is the sum of all words. There is no minimum or maximum score, whereas more words indicate a better outcome.
  During the CFT test, the subject is given 1 minute to produce as many unique words as possible within a semantic category. The subject's score is the number of unique correct words.
  There is no minimum or maximum score whereas a score of under 14 is interpreted as concerning regarding cognition.
Time Frame: Baseline, Week 12
Population: Total NTB score is the sum of 'Total correct response' of Category Fluency Test (CFT) and 'Total number of correct words' of Controlled Oral Word Association Test (COWAT). Each score ('Total correct response' of CFT and 'Total number of correct word' of COWAT) will also be analysed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xanamem™ | Placebo
Number analyzed (Participants) | 86 | 91
score on a scale
  COWAT Total Correct Words | 0.5 (8.08) | 0.5 (8.12)
  CTF Total Correct Responses | 0.3 (8.53) | -0.7 (6.28)
  NTB Total Score | 0.8 (11.50) | -0.2 (9.84)

8. Other Pre Specified Outcome: Pregnancy Test
Description: Women of childbearing potential only. Serum pregnancy test at screening and a urine pregnancy test at all subsequent clinic visits
Time Frame: Screening, baseline, Week 4, Week, 8, Week 12, Week 16
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Optional PD Assessment - Changes in Pharmacodynamic (PD) Measures of Testosterone
Description: This assessment will be carried out on subjects who consented to this optional test. PD sample will be collected at pre-dose at each required visit
Time Frame: Screening, baseline, Week 4, Week, 8, Week 12, Week 16
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Optional PD Assessment - Changes in Pharmacodynamic (PD) Measures of Androstenedione
Description: as for outcome 9
Time Frame: Screening, baseline, Week 4, Week, 8, Week 12, Week 16
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Optional PD Assessment - Changes in Pharmacodynamic (PD) Measures of Dehydroepiandrosterone Sulfate (DHEAS)
Description: as for outcome 9
Time Frame: Screening, baseline, Week 4, Week, 8, Week 12, Week 16
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Optional PD Assessment - Changes in Pharmacodynamic (PD) Measures of Adrenocorticotropic Hormone (ACTH)
Description: as for outcome 9
Time Frame: Screening, baseline, Week 4, Week, 8, Week 12, Week 16
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Pharmacokinetics (PK), Including Analysis of Cortisol Levels
Description: as for outcome 9
Time Frame: Baseline, Week 4, Week 8, Week 12 and Unscheduled Safety Visit
Reporting Status: Not Posted

14. Other Pre Specified Outcome: NTSS-6
Description: Change in Neuropathy Total Symptom Score (NTSS-6)
Time Frame: Screening, Baseline, Week 4, Week 8, Week 12, Week 16, Ad Hoc and Unscheduled Safety Visit
Reporting Status: Not Posted

15. Other Pre Specified Outcome: NFM
Description: Change in Nerve Function Monitoring (NFM)
Time Frame: Screening, Baseline, Week 4, Week 8, Week 12, Week 16
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Vital Signs
Description: Change in Vital Signs (including Heart Rate, Blood Pressure, Body Weight, BMI)
Time Frame: Screening, Baseline, Week 4, Week 8, Week 12, Week 16, Unscheduled Safety Visit
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Metabolic Function
Description: Change in Metabolic Function Test Results of Lipids, Glucose, Hemoglobin A1c (HbA1c)
Time Frame: Baseline, Week 12
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Clinical Safety Laboratory Values
Description: Change in Clinical Safety Laboratory Values (biochemistry, hematology, urine examination)
Time Frame: Screening, Baseline, Week 4, Week 8, Week 12, Week 16
Reporting Status: Not Posted

19. Other Pre Specified Outcome: AEs
Description: Incidence of Adverse Events (AEs)
Time Frame: Screening, Baseline, Week 4, Week 8, Week 12, Week 16, Ad Hoc
Reporting Status: Not Posted

20. Other Pre Specified Outcome: ECG
Description: Change in Electrocardiogram (ECG) Values
Time Frame: Screening, Baseline, Week 4, Week 8, Week 12, Week 16
Reporting Status: Not Posted

21. Other Pre Specified Outcome: CSSRS
Description: Change in Scores of Columbia Suicide Severity Rating Scale (CSSRS)
Time Frame: Screening, Week 4, Week 8, Week 12, Week 16
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Median treatment duration (weeks) was 12 weeks (range: 0.14, 13.0 weeks) for subjects in the Xanamem group and 12 weeks (range: 0.14, 13.1 weeks) for subjects in the placebo group.
Arm/Group | Xanamem™ | Placebo
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/94
Serious Adverse Events (participants affected / at risk) | 4/91 | 4/94
Other Adverse Events (participants affected / at risk) | 33/91 | 32/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xanamem™ (N=91) | Placebo (N=94)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Vibration test abnormal (Investigations) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Pulmonary Cavitation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xanamem™ (N=91) | Placebo (N=94)
Headache (Nervous system disorders) | 9 | 10
Urinary tract infection (Infections and infestations) | 6 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Fall (Injury, poisoning and procedural complications) | 3 | 6
Dizziness (Nervous system disorders) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT02727699/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT02727699/SAP_002.pdf